CLINICAL TRIAL: NCT00975572
Title: A Double-blind, Randomized, Stratified and Controlled Clinical Trial With Split-virion, Adjuvanted and Non-adjuvanted Influenza A/H1N1 Vaccines in Healthy Adults, Elders, Adolescents and Children
Brief Title: Novel Influenza A/H1N1 Split- Virion Vaccine in Healthy Population Aged 3 Years and Older
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Hualan Biological Bacterin Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Fengcai Zhu, Prof., Jiangsu Province Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JSVCT001
Record Dates: First submitted 2009-09-08; First posted 2009-09-11 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2009-09

CONDITIONS: Virus Diseases; Respiratory Tract Diseases; Respiratory Tract Infections; Influenza; Orthomyxoviridae Infections
Keywords: Flu; adjuvanted H1N1 vaccine; non-adjuvanted H1N1 vaccine; Immunogenictiy; Safety
MeSH Terms: conditions — Virus Diseases; Respiratory Tract Diseases; Respiratory Tract Infections; Influenza, Human; Orthomyxoviridae Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- split-virion, adjuvanted H1N1 vaccine of 7.5 μg (Experimental)
  Interventions: Biological: Experimental: split-virion, adjuvanted H1N1 vaccine of 7.5 μg
- split-virion, adjuvanted H1N1 vaccine of 15 μg (Experimental)
  Interventions: Biological: Experimental: split-virion, adjuvanted H1N1 vaccine of 15 μg
- split-virion, adjuvanted H1N1 vaccine of 30 μg (Experimental)
  Interventions: Biological: Experimental: split-virion, adjuvanted H1N1 vaccine of 30 μg
- split-virion, non-adjuvanted H1N1 vaccine of 15 μg (Experimental)
  Interventions: Biological: Experimental: split-virion, non-adjuvanted H1N1 vaccine of 15 μg
- Placebo control (Placebo Comparator)
  Interventions: Biological: Placebo Comparator: Placebo control
- split-virion, non-adjuvanted H1N1 vaccine of 30 μg (Experimental)
  Interventions: Biological: split-virion, non-adjuvanted H1N1 vaccine of 30 μg

INTERVENTIONS:
Biological: split-virion, non-adjuvanted H1N1 vaccine of 30 μg — 440 participants (110 elders, 110 adults, 110 adolescents and 110 children) to receive split-virion, non-adjuvanted H1N1 vaccine of 30 μg on day 0 and 21.
  Arms: split-virion, non-adjuvanted H1N1 vaccine of 30 μg
Biological: Experimental: split-virion, adjuvanted H1N1 vaccine of 7.5 μg — 440 participants (110 elders,110 adults, 110 adolescents and 110 children) to receive split-virion, adjuvanted H1N1 vaccine of 7.5 μg on day 0 and 21.
  Arms: split-virion, adjuvanted H1N1 vaccine of 7.5 μg
Biological: Experimental: split-virion, adjuvanted H1N1 vaccine of 15 μg — 440 participants (110 elders, 110 adults, 110 adolescents and 110 children) to receive split-virion, adjuvanted H1N1 vaccine of 15 μg on day 0 and 21.
  Arms: split-virion, adjuvanted H1N1 vaccine of 15 μg
Biological: Experimental: split-virion, adjuvanted H1N1 vaccine of 30 μg — 330 participants (110 elders, 110 adults, and 110 adolescents) to receive split-virion, adjuvanted H1N1 vaccine of 30 μg on day 0 and 21.
  Arms: split-virion, adjuvanted H1N1 vaccine of 30 μg
Biological: Experimental: split-virion, non-adjuvanted H1N1 vaccine of 15 μg — 440 participants (110 elders, 110 adults, 110 adolescents and 110 children) to receive split-virion, non-adjuvanted H1N1 vaccine of 15 μg on day 0 and 21.
  Arms: split-virion, non-adjuvanted H1N1 vaccine of 15 μg
Biological: Placebo Comparator: Placebo control — 110 adults to receive placebo control (Phosphate Buffer Saline) on day 0 and 21.
  Arms: Placebo control

SUMMARY:
The primary safety objective of this study is to assess the safety of split- virion inactivated H1N1 vaccine with and without adjuvant when administered at the 7.5,15 or 30 mcg dose. The primary immunogenicity objective is to assess the antibody response following each dose of split- virion inactivated A(H1N1) vaccine with and without adjuvant. Participants will include up to 2200 healthy persons age 3 and older who have no history of novel influenza H1N1 2009 infection or novel influenza H1N1 2009 vaccination. This is a randomized, double-blinded, Phase II study in healthy males and non-pregnant females, aged 3 years and older. Subjects will be stratified by elders (equal to or more than 61 years), adults (18-60 years), adolescents (12-17 years) and children (3-11 years), elders and adolescents will be randomized into 5 dose groups (adjuvanted H1N1 vaccine of 7.5,15 or 30 mcg per dose or non-adjuvanted H1N1 vaccine of 15 or 30 mcg per dose), children will be randomized into 4 dose groups (adjuvanted H1N1 vaccine of 7.5 or 15 mcg per dose or non-adjuvanted H1N1 vaccine of 15 or 30 mcg per dose), adults will be randomized into 6 dose groups (adjuvanted H1N1 vaccine of 7.5,15 or 30 mcg per dose or non-adjuvanted H1N1 vaccine of 15 or 30 mcg per dose or placebo), 110 subjects per dose and age stratum will be to receive intramuscular influenza H1N1 vaccine. The H1N1 vaccine will be administered at Day 0 and Day 21. Following immunization, safety will be measured by assessment of adverse events through 21 days following the last vaccination (Day 42 for those receiving both doses), serious adverse events and new-onset chronic medical conditions through 6 months post the final vaccination (Day 180 after second vaccination), and reactogenicity to the vaccine for 8 days (Day 0-7) following each vaccination. Immunogenicity testing will be hemagglutination inhibiting (HAI) on serum obtained on the day 21 of each vaccination (prior to vaccination), on Day 21 after first vaccination, and 21 days following the second vaccination (Day 42).

DETAILED DESCRIPTION:
Recently, a novel swine-origin influenza A/H1N1 virus was identified as a significant cause of febrile respiratory illnesses in Mexico and the United States. It rapidly spread to many countries around the world, prompting the World Health Organization (WHO) to declare a pandemic on June 11, 2009. Data from several cohorts in different age groups that received licensed trivalent seasonal influenza vaccines suggest that these vaccines are unlikely to provide protection against the new virus. In addition, adults are more likely to have measurable levels of serum hemagglutination inhibition assay (HAI) or neutralizing antibody than are children. These data indicate the need to develop vaccines against the new H1N1 strain and suggest that different vaccine strategies (e.g., number of doses, need for adjuvant) may be appropriate for persons in different age groups. The primary safety objective of this study is to assess the safety of split- virion inactivated H1N1 vaccine with and without adjuvant when administered at the 7.5,15 or 30 mcg dose. The primary immunogenicity objective is to assess the antibody response following each dose of split- virion inactivated A(H1N1) vaccine with and without adjuvant,. Participants will include up to 2200 healthy persons age 3 and older who have no history of novel influenza H1N1 2009 infection or novel influenza H1N1 2009 vaccination. This is a randomized, double-blinded, Phase II study in healthy males and non-pregnant females, aged 3 years and older. This study is designed to investigate the safety, reactogenicity, and immunogenicity of an inactivated influenza H1N1 virus vaccine at different dose levels of split- virion inactivated H1N1 vaccine with or without adjuvant or placebo in 4 aged groups. Subjects will be stratified by elders (equal to or more than 61 years), adults (18-60 years), adolescents (12-17 years) and children (3-11 years), elders and adolescents will be randomized into 5 dose groups(adjuvanted H1N1 vaccine of 7.5,15 or 30 mcg per dose or non-adjuvanted H1N1 vaccine of 15 or 30 mcg per dose ) , children will be randomized into 4 dose groups(adjuvanted H1N1 vaccine of 7.5 or 15 mcg per dose or non-adjuvanted H1N1 vaccine of 15 or 30 mcg per dose ), adults will be randomized into 6 dose groups(adjuvanted H1N1 vaccine of 7.5,15 or 30 mcg per dose or non-adjuvanted H1N1 vaccine of 15 or 30 mcg per dose or placebo ), 110 subjects per dose and age stratum will be to receive intramuscular influenza H1N1 vaccine . The H1N1 vaccine will be administered at Day 0 and Day 21. Following immunization, safety will be measured by assessment of adverse events through 21 days following the last vaccination (Day 42 for those receiving both doses), serious adverse events and new-onset chronic medical conditions through 6 months post the final vaccination (Day 180 after second vaccination), and reactogenicity to the vaccine for 8 days (Day 0-7) following each vaccination. Immunogenicity testing will be HAI on serum obtained on the day 21 of each vaccination (prior to vaccination), on Day 21 after first vaccination, and 21 days following the second vaccination (Day 42).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female aged 3 and older
2. Be able to show legal identity card for the sake of recruitment
3. Volunteers or their guardians are able to understand and sign the informed consent

Exclusion Criteria:

1. Cases, cured cases and close contact of influenza A (H1N1) virus
2. Women of pregnancy, lactation or about to be pregnant in 60 days
3. Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine, such as egg, egg protein, etc
4. Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
5. Autoimmune disease or immunodeficiency
6. Asthma that is unstable or required emergent care, hospitalization or intubation during the past two years or that required the use of oral or intravenous corticosteroids
7. Diabetes mellitus (type I or II), with the exception of gestational diabetes
8. History of thyroidectomy or thyroid disease that required medication within the past 12 months
9. Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years
10. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
11. Active malignancy or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of study
12. Seizure disorder other than:

    * Febrile seizures under the age of two years old
    * Seizures secondary to alcohol withdrawal more than 3 years ago, or
    * A singular seizure not requiring treatment within the last 3 years
13. Asplenia, functional asplenia or any condition resulting in the absence or removal o the spleen
14. Guillain-Barre Syndrome
15. Any history of immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis)
16. History of any blood products or seasonal influenza vaccine administration within 3 months before the dosing
17. Administration of any other investigational research agents within 30 days before the dosing
18. Administration of any live attenuated vaccine within 30 days before the dosing
19. Administration of subunit or inactivated vaccines, e.g., pneumococcal vaccine, or allergy treatment with antigen injections, within 14 days before the dosing
20. Be receiving anti-TB prophylaxis or therapy currently
21. Axillary temperature > 37.0 centigrade at the time of dosing
22. Psychiatric condition that precludes compliance with the protocol:

    * Past or present psychoses
    * Past or present bipolar disorder requiring therapy that has not been well controlled on medication for the past two years
    * Disorder requiring lithium
    * Suicidal ideation occurring within five years prior to enrollment
23. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent

Ages: 3 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2200 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Hemagglutination inhibition antibody titer | D0,D21,D35

SECONDARY OUTCOMES:
local and systemic adverse reaction after vaccination | D0-42

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Cai Zhu, Master, Principal Investigator — Jiangsu CDPC
Locations (1):
- Taizhou Municipal Center for Disease Control and Prevention, Taizhou, Jiangsu, China

REFERENCES:
- [Derived] Liang XF, Wang HQ, Wang JZ, Fang HH, Wu J, Zhu FC, Li RC, Xia SL, Zhao YL, Li FJ, Yan SH, Yin WD, An K, Feng DJ, Cui XL, Qi FC, Ju CJ, Zhang YH, Guo ZJ, Chen PY, Chen Z, Yan KM, Wang Y. Safety and immunogenicity of 2009 pandemic influenza A H1N1 vaccines in China: a multicentre, double-blind, randomised, placebo-controlled trial. Lancet. 2010 Jan 2;375(9708):56-66. doi: 10.1016/S0140-6736(09)62003-1. Epub 2009 Dec 15. PMID 20018364
- [Derived] Zhu FC, Wang H, Fang HH, Yang JG, Lin XJ, Liang XF, Zhang XF, Pan HX, Meng FY, Hu YM, Liu WD, Li CG, Li W, Zhang X, Hu JM, Peng WB, Yang BP, Xi P, Wang HQ, Zheng JS. A novel influenza A (H1N1) vaccine in various age groups. N Engl J Med. 2009 Dec 17;361(25):2414-23. doi: 10.1056/NEJMoa0908535. Epub 2009 Oct 21. PMID 19846844